CLINICAL TRIAL: NCT00392808
Title: Randomized, Open Label, Active Control, Parallel Assignment Clinical Trial to Evaluate the Immunogenicity of Polysaccharide Meningococcal C Vaccines Conjugated With Tetanus Toxoid or CRM197 Given as a Booster Dose at 14-18 Months of Life.
Brief Title: Immunogenicity of the Booster Dose of Two MenC Vaccines
Acronym: CSISP-MENC1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Superior de Investigación en Salud Publica (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSISP-VAC-MENC1; EUDRA 2006-003525-82
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Results first posted 2013-10-11 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-08

CONDITIONS: Meningococcal Infection
Keywords: Meningococcal vaccine; Immunization, secondary; vaccines conjugated; Meningococcal disease
MeSH Terms: conditions — Meningococcal Infections; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- MENC-CRM/MENC-CRM (Experimental): Children primed with 3 doses of MenC-CRM vaccine, Intervention: boosted with one dose of MenC-CRM vaccine
  Interventions: Biological: conjugated polysaccharide menC vaccine
- MENC-CRM/MENC-TT (Experimental): Children Primed with three doses of MenC-CRM vaccine. Intervention: boosted with one dose of MenC-TT
  Interventions: Biological: conjugated polysaccharide menC vaccine
- MENC-TT/MENC-CRM (Experimental): Children primovacccinated with two MenC-TT vaccine doses. Intervention: boosted with one dose MenC-CRM vaccine
  Interventions: Biological: conjugated polysaccharide menC vaccine
- MENC-TT/MENC-TT (Experimental): Children primovacccinated with two MenC-TT vaccine doses. Intervention boosted with one dose MenC-TT vaccine
  Interventions: Biological: conjugated polysaccharide menC vaccine

INTERVENTIONS:
Biological: conjugated polysaccharide menC vaccine — Booster vaccine dose at 14 to 18 months.

SUMMARY:
The purpose of the study is to evaluate the immune response of toddlers, to a booster dose in the second year of life of two meningococcal C conjugated polysaccharide vaccine, and to assess the interchangeability of the two different vaccines.

DETAILED DESCRIPTION:
Children 14 to 18 months of life, previously vaccinated with 2 doses of tetanus toxoid conjugated polysaccharide men C vaccine or three doses of the CRM197 conjugated polysaccharide men C vaccine before 7 months of age, are randomized to receive any of the two vaccines. Serum antibody activity against meningococcus C will be measured inmediately before and 4 weeks after the booster dose. Children will also be vaccinated with a combined vaccine containing DTaP+IPV+Hib.

ELIGIBILITY:
Inclusion Criteria:

* Healthy toddlers of both sexes
* Toddlers of 14 to 19 months of age (including the day that the toddler is 14 and the day before he is 19 months of age)
* Children previously vaccinated with two doses of polysaccharide meningococcal C vaccine conjugated to tetanus toxoid or three doses of polysaccharide meningococcal C conjugated to CRM197 before 7 month of age.
* Informed consent signed by one or both parents who are adequately informed about the study.

Exclusion Criteria:

* Toddlers with severe diseases or axilar temperature ≥ 38,0ºC at inclusion time
* Toddlers with severe chronic diseases
* Toddlers who have received any other vaccine within the last month or with a programmed vaccination within the 28 subsequent days after the administration of the vaccine of study.
* Toddlers with clinical or bacteriological diagnosis of previous meningococcal disease.
* Toddlers with hypersensitivity to any of the components of the vaccines to study or antibiotics used during the manufacturing process that could be present as non- detectable traces (streptomycin, neomycin, polymyxin B).
* Toddlers with personal history of convulsions.
* Toddlers with known bleeding disorder no controlled
* Toddlers with known congenital or acquired immunodeficiency
* Toddlers who are receiving or have been received any treatment that could change the immune response (administration of intravenous immunoglobulin, systemic corticosteroids or haemoderivates) within the 3 previous months.
* A toddler that under investigator opinion is probable to be lost during the follow-up
* A toddler that is currently included or is planned to be included in any other clinical trial.
* A toddler that under investigator opinion must not be included in the study due to other medical or social reasons.

Ages: 14 Months to 19 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 389 (Actual)
Dates: Start 2007-01; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Diez-Domingo, PhD, Study Chair — Centro Superior Investigacion Salud Publica (CSISP)
Locations (2):
- Spain (2):
  - Universidad Rey Juan Carlos I, Madrid
  - Centro Superior Investigación en Salud Publica, Valencia

REFERENCES:
- [Result] Diez-Domingo J, Planelles-Cantarino MV, Baldo-Torrenti JM, Ubeda-Sansano I, Jubert-Rosich A, Puig-Barbera J, Gutierrez-Gimeno MV. Antibody persistence 12 months after a booster dose of meningococcal-C conjugated vaccine in the second year of life. Pediatr Infect Dis J. 2010 Aug;29(8):768-70. doi: 10.1097/INF.0b013e3181d9e653. PMID 20375851
- [Result] Diez-Domingo J, Cantarino MV, Torrenti JM, Sansano MI, Rosich AJ, Merino AH, de Miguel AG, Gonzalez JB, Marcos MD; MenC Study Group. A randomized, multicenter, open-label clinical trial to assess the immunogenicity of a meningococcal C vaccine booster dose administered to children aged 14 to 18 months. Pediatr Infect Dis J. 2010 Feb;29(2):148-52. doi: 10.1097/INF.0b013e3181b9a831. PMID 19927040

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was done in primary care pediatric clinics, between january and may 2007.
Groups:
- MENC-TT/MENC-TT: Children primovacccinated with two MenC-TT vaccine doses and primed with MenC-TT vaccine
- MENC-TT/MENC-CRM: Children primovacccinated with two MenC-TT vaccine doses and primed with MenC-CRM vaccine
- MENC-CRM/MENC-TT: Children Primed with three doses of MenC-CRM vaccine and boosted with MenC-TT
- MENC-CRM/MENC-CRM: Children primed with 3 doses of MenC-CRM vaccine, and boosted with MenC-CRM vaccine
Period: Overall Study
Arm/Group | MENC-TT/MENC-TT | MENC-TT/MENC-CRM | MENC-CRM/MENC-TT | MENC-CRM/MENC-CRM
Started | 87 | 89 | 109 | 104
Completed | 81 | 86 | 107 | 100
Not Completed | 6 | 3 | 2 | 4
Not completed — Lost to Follow-up | 3 | 2 | 1 | 2
Not completed — Unable to withdraw blood | 3 | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MENC-CRM/MENC-CRM | MENC-CRM/MENC-TT | MENC-TT/MENC-CRM | MENC-TT/MENC-TT | Total
Number analyzed (Participants) | 104 | 109 | 89 | 87 | 389
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 104 | 109 | 89 | 87 | 389
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 1.37 (0.23) | 1.38 (0.13) | 1.43 (0.23) | 1.46 (0.09) | 1.4 (.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 53 | 46 | 45 | 202
  Male | 46 | 56 | 43 | 42 | 187
Region of Enrollment [Number; unit: participants]
  Spain | 104 | 109 | 89 | 87 | 389

OUTCOME MEASURES:

1. Primary Outcome: Serum Bactericidal Activity Against MenC
Time Frame: One month after booster dose
Measure: Geometric Mean (95% Confidence Interval); unit: GMTs
Arm/Group | MENC-TT/MENC-TT | MENC-TT/MENC-CRM | MENC-CRM/MENC-TT | MENC-CRM/MENC-CRM
Number analyzed (Participants) | 81 | 86 | 107 | 100
GMTs | 6786 [5023 to 9167] | 6278 [5359 to 7932] | 2061 [1599 to 2627] | 1746 [1378 to 2213]

2. Primary Outcome: Serum Antibody Titers Against Haemophilus Influenzae Type b.
Time Frame: One year
Measure: Geometric Mean (95% Confidence Interval); unit: GMCs
Arm/Group | MENC-TT/MENC-TT | MENC-TT/MENC-CRM | MENC-CRM/MENC-TT | MENC-CRM/MENC-CRM
Number analyzed (Participants) | 76 | 79 | 83 | 79
GMCs | 23.8 [17.5 to 32.4] | 30.8 [23.7 to 40.1] | 30.5 [23.3 to 40.0] | 26.0 [19.1 to 35.4]

ADVERSE EVENTS:
Arm/Group | MENC-TT/MENC-TT | MENC-TT/MENC-CRM | MENC-CRM/MENC-TT | MENC-CRM/MENC-CRM
Serious Adverse Events (participants affected / at risk) | 3/87 | 5/89 | 2/109 | 2/104
Other Adverse Events (participants affected / at risk) | 0/87 | 1/89 | 6/109 | 5/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MENC-TT/MENC-TT (N=87) | MENC-TT/MENC-CRM (N=89) | MENC-CRM/MENC-TT (N=109) | MENC-CRM/MENC-CRM (N=104)
Febrile seizures (Nervous system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
cutaneous abscess (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leishmaniasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
asthma (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MENC-TT/MENC-TT (N=87) | MENC-TT/MENC-CRM (N=89) | MENC-CRM/MENC-TT (N=109) | MENC-CRM/MENC-CRM (N=104)
local reactions: pain, induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 5 (5) | 5 (5)
fever (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
acropustulosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes